CLINICAL TRIAL: NCT01138878
Title: HIV Testing in Non-traditional Settings Study
Acronym: HINTS
Status: Completed | Type: Observational
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Collaborators: Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government); Public Health England (Other Government); Homerton University Hospital NHS Foundation Trust (Other); King's College Hospital NHS Trust (Other); Hammersmith and Fulham Primary Care Trust (Unknown)
Responsible Party: Dr Ann Sullivan, Chelsea and Westminster NHS Foundation Trust
Other Study IDs: 1.4
Record Dates: First submitted 2010-06-04; First posted 2010-06-08 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2010-05

CONDITIONS: HIV
Keywords: HIV; testing; non traditional settings; acceptability; feasibility
MeSH Terms: interventions — Surveys and Questionnaires; HIV Testing

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Patient pre-study group: A set of all 16-65 yr olds (not know already to be HIV-positive) accessing the healthcare setting prior to the introduction of the HIV testing pilot programme
  Interventions: Other: Questionnaire; Other: Focus Group Discussion
- Staff pre-study group: A set of staff working within the healthcare setting prior to the introduction of the HIV screening programme
  Interventions: Other: Questionnaire; Other: Focus Group Discussion
- Patient intra-study group: A set of patients, aged 16-65 and known not to be HIV-positive, who access the healthcare setting during the HIV testing pilot programme
  Interventions: Other: Questionnaire; Other: HIV test (serum or salivary); Other: Semi-structured telephone interview
- Post-study staff group: A set of staff who worked within the healthcare setting for the duration of the HIV testing pilot programme
  Interventions: Other: Questionnaire; Other: Focus Group Discussion

INTERVENTIONS:
Other: Questionnaire — Administration of written questionnaire to assess attitudes towards the introduction of routine HIV testing programmes to that healthcare setting
Other: Focus Group Discussion — FGD to explore attitudes within each group towards the introduction of routine HIV screening programmes in each medical setting
  Groups: Patient pre-study group; Post-study staff group; Staff pre-study group
Other: HIV test (serum or salivary) — An HIV test offered to all 16-65 year olds (not known already to be HIV-positive) accessing the healthcare setting during the twelve week pilot period
  Groups: Patient intra-study group
Other: Semi-structured telephone interview — Telephone interview administered to patients offered an HIV test during the pilot period
  Groups: Patient intra-study group

SUMMARY:
Surveillance data suggests that approximately one third of the 82 000 HIV infected adults in the UK remain undiagnosed - that is, they are living with the infection but do not know this. The majority of HIV testing in the UK to date has taken place in sexual health clinics and in antenatal care. Published National guidelines advocate routine HIV testing of 16-65 year olds in more general healthcare settings in parts of the country with relatively high rates of HIV (more than 2 per thousand individuals diagnosed locally). The HINTS Study investigates the utility, feasibility and acceptability, to patients and staff, of offering routine HIV testing in four general medical settings, all set in areas of high HIV prevalence. The settings comprise: Primary Care, Outpatients, an Acute Care Unit and an Emergency Department.

ELIGIBILITY:
Inclusion Criteria (patient study only):

* aged 16 - 65 and accessing relevant healthcare setting for care
* able to consent to HIV test
* able to provide adequate contact details
* to complete written questionnaire: adequate written English
* to participate in focus group discussion (pre-study group)/participate in semi-structured telephone interview (intra-study group): ability to provide fully informed consent

Exclusion Criteria:

* known HIV positive
* unable to provide adequate contact details
* unable to provide consent (to HIV test and/or participation in questionnaire/focus group/semi-structured interview studies)

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: For patient pre-study and intra-study: All patients aged 16-65 (not know already to be HIV positive) attending the healthcare setting (Primary Care centre, Emergency Department, Acute Care Unit, Medical Outpatient Clinic) before or during the twelve week HIV testing pilot programme
  For Staff pre-study and post-study: All members of staff (HCP, Allied Health Professionals and Admin/Clerical) working within the healthcare settings examined before and during the implementation of the HIV testing programme
Sampling Method: Non-Probability Sample
Enrollment: 6350 (Actual)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
(1) Feasibility of delivering opt-out HIV testing in ED/ACU/OPD/Primary Care setting | At end of twelve week testing period at each site

SECONDARY OUTCOMES:
(2) Estimate of prevalence of undiagnosed HIV with risk factor/demographic assessment | At end of twelve week testing period

CONTACTS AND LOCATIONS:
Overall Officials: Ann K Sullivan, MBBS FRCP, Principal Investigator — Chelsea and Westminster NHS Foundation Trust; Jane Anderson, MBBS FRCP, Principal Investigator — Homerton University Hospital NHS Foundation Trust; Melinda Tenant-Flowers, MBBS FRCP MSc, Principal Investigator — Kings College Hospital NHS Foundation Trust
Locations (4):
- United Kingdom (4):
  - Homerton University NHS Foundation Trust, London
  - Kings College Hospital NHS Foundation Trust, London
  - Chelsea and Westminster NHS Foundation Trust, London
  - North End Medical Centre, Hammersmith and Fulham Primary Care NHS Trust, London